CLINICAL TRIAL: NCT02276781
Title: BRAVO: Biomarker Risk Assessment in Vulnerable Outpatients
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine, Northwestern University
Other Study IDs: R01HL089619 (NIH); R01HL089619 (NIH)
Record Dates: First submitted 2014-10-24; First posted 2014-10-28 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; Peripheral Arterial Disease; Biomarkers
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: EDTA plasma, Citrate plasma, serum, whole blood (DNA)* and RNA*. Lower extremity muscle biopsies*
  *genetic factors and muscle biopsies are optional study elements
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PAD Participants: PAD participants from among consecutive patients with PAD identified from Chicago area non-invasive vascular laboratories

SUMMARY:
The investigators hypothesize that among people with lower extremity peripheral artery disease (PAD), biomarker levels are higher during time periods immediately preceding an acute coronary event compared to time periods not immediately preceding an acute coronary event. Biomarkers the investigators will study are CRP, SAA, and D-dimer. Biomarkers will be measured at baseline and every two months during follow-up.

The primary aims of this study are as follows. Specific Aim #1. Among participants with PAD who experience an acute coronary event during follow-up, the investigators will determine whether biomarker levels measured immediately prior to the coronary event are higher than levels that do not immediately precede coronary events. Specific Aim #2, Part 1. The investigators will determine whether participants who experience a coronary event (cases) have higher biomarker levels at the visit immediately prior to the event than participants who have not experienced a coronary event (controls) at the time of the case event. Specific Aim #2, Part 2. The investigators will determine whether participants who experience a coronary event (cases) have a greater increase in biomarkers during the time period leading up to the event compared to participants who have not experienced a coronary event (controls).

To achieve these aims, the investigators will enroll up to 650 participants with PAD and follow them prospectively, measuring blood samples every two months, and ascertaining the presence of acute coronary events every two months.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arterial disease defined as an ABI less than or equal to 0.90 in either leg

We will also include PAD patients with an ABI > 0.90 who meet any of the following criteria:

* History of documented lower extremity revascularization. A written report from the medical record will be required as documentation
* An angiogram demonstrating >50% stenosis in one or more lower extremity arteries. Again, a written report will be required to document this. Participants with an angiogram noting moderate or greater stenosis will also be considered eligible, when a specific amount of stenosis is not denoted
* A report from the non-invasive vascular laboratory demonstrating a toe brachial pressure less than 0.60. Other criteria (i.e. PVR data) from the non-invasive vascular laboratory will not be considered sufficient for inclusion

Exclusion Criteria:

* Treatment for cancer other than non-melanoma skin cancer during the previous 2 years. (However, persons treated for non-invasive breast cancer or prostate cancer during the previous year will be potentially eligible if their physician indicates that their life expectancy is > 24 months, since non-invasive breast and prostate cancer often have an excellent prognosis)
* Unintentional weight loss of > 7.5 pounds in the last six months;
* Mini-Mental Status Exam (MMSE) score < 23 out of 30 or other history of cognitive impairment
* Communication difficulty due to language barriers
* Refusal to have regular blood draws or inability to obtain a blood sample at baseline
* Coronary or cerebrovascular event during the previous six months (these persons may become eligible at a later date)
* History of inflammatory arthritis (rheumatoid arthritis, lupus erythematosis, or polymyalgia rheumatic, gout), however participants with gouty arthritis will be eligible if the last episode was more than three months ago
* Residence more than 40 miles away from the medical center and unwillingness to travel to the medical center for every two month blood collection
* Unable to return for follow up testing for > a consecutive six month period in the next two years
* Heart transplant surgery
* Major surgery (one that required general anesthesia) within the past 3 months These persons may become eligible at a later date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PAD participants from among consecutive patients with PAD identified from Chicago area non-invasive vascular laboratories and vascular surgery, cardiology, general internal medicine, geriatric, and endocrinology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
fatal and non-fatal coronary events | Every two months for up to three and a half years
  Our primary outcome is fatal and non-fatal coronary events. Non-fatal coronary events will be defined as acute myocardial infarction (MI), hospitalizations for unstable angina, and new ECG findings consistent with MI

CONTACTS AND LOCATIONS:
Overall Officials: Mary M McDermott, MD, Principal Investigator — Northwestern University
Locations (6):
- United States (6):
  - Mt. Sinai Medical Center, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Jesse Brown Veterans Administration Medical Center, Chicago, Illinois
  - Rush Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - St. Joseph's Hospital, Chicago, Illinois